CLINICAL TRIAL: NCT02292095
Title: Effects of Transverse Abdominis Plane Block Guided by Ultrasound on the Postoperative Analgesia and Quality of Lives Among the Patients Undergo Inguinal Hernia Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, The Department of Anestheiology and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYYMZ-002
Record Dates: First submitted 2014-11-08; First posted 2014-11-17 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Post-operative Pain; Inguinal Hernia
Keywords: anesthesia; transverse abdominis plane block; patient controlled intravenous analgesia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAPB group (Experimental): Participants in this group will receive transverse abdominis plane block combined with patient controlled intravenous analgesia.Transverse abdominis plane block will be guided by ultrasound and 0.75% 20 ml ropivacaine will be injected with the sonographic view at the end of the surgery.Participants in this group will also receive patient controlled intravenous analgesia after surgery,the regimens of patient controlled intravenous analgesia are included tramadol 800 mg, flurbiprofenaxetil 100 mg, and dexamethasone 5 mg with saline added up to a volume of 80 ml in total
  Interventions: Procedure: TAPB group
- PCIA group (Active Comparator): Participants in this group will only receive patient controlled intravenous analgesia after surgery.The formula of the PCIA included tramadol 800 mg, flurbiprofenaxetil 100 mg, and dexamethasone 5 mg with saline added up to a volume of 80 ml in total, they received a loading dose of 2 ml followed by an infusion rate of 1 ml/h with bolus of 2 ml, the lock time was set at 15 min
  Interventions: Procedure: PCIA group

INTERVENTIONS:
Procedure: TAPB group — transverse abdominis plane block will be conducted by ultrasound and a single-injection of 20ml 0.75% ropivacaine will be conducted for nerve block at the end of surgery.After surgery,participants in this group will also receive patient controlled intravenous analgesia.
  Arms: TAPB group
Procedure: PCIA group — The formula of patient controlled intravenous analgesia included tramadol 800 mg, flurbiprofenaxetil 100 mg, and dexamethasone 5 mg with saline added up to a volume of 80 ml in total, they received a loading dose of 2 ml followed by an infusion rate of 1 ml/h with bolus of 2 ml, the lock time was set at 15 min
  Arms: PCIA group

SUMMARY:
The incidence of post-operative pain after open inguinal hernia repair is high and impair the quality of lives of the patients.The purpose of this study is to determine whether transverse abdominis plane block combined with intravenous patient controlled analgesia is superior to intravenous patient controlled analgesia in improving the quality of life and reducing the incidence of chronic post-surgical pain

DETAILED DESCRIPTION:
The incidence of post-operative pain after open inguinal hernia repair is high according to a a larger-sample epidemic research. Meanwhile, the investigators also found the incidence of CPSP of herniorrhaphy was 37.8% among the patients with PCA, and the incidence of neuropathic pain was 37.5% in these patients with CPSP. European hernia society has proposed that local infiltration anesthesia was suggested to all patients without any contraindications who undergo inguinal hernia repair. Transverse abdominis plane block(TABP),which injecting local anesthetics into the interval between obliquus internus abdominis muscle and transverse abdominal muscle could block the abdominal nerve and could alleviate the pain postoperatively. TABP can block the two mainly nerve (iliohypogastric nerve, ilioinguinal nerve) for inguinal hernia repair and so it seems to have a good effects to relieve the pain of inguinal hernia repair. So the investigators conduct the randomized controlled trial to investigate whether transversus abdominis plane block combined with intravenous patient controlled analgesia is superior to intravenous patient controlled analgesia in improving the quality of life and reducing the incidence of chronic post-surgical pain.

This study was approved by the Medical Ethics Committee of the First Affiliated Hospital of Chongqing Medical University. All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study. This study is a prospective, randomized, controlled clinical trial guided by the standard of good clinical practice (GCP), and eligible participants are divided into two groups: group TAPB and group PCIA, and assess the outcomes of the incidence of acute and chronic postoperative pain and the effects of the two methods on the quality of lives of patients undergo inguinal hernia repair.

Participants in group TAPB will receive transversus abdominis plane block guided by ultrasound at the end of the surgery and also receive intravenous patient controlled analgesia after surgery.

Participants in group PCIA will only receive intravenous patient controlled analgesia after surgery.

The primary outcome of the study is VAS scores at rest and in motion at 3 months postoperatively. The secondary outcomes of this study are chronic post-surgical pain at 6 and 12 months postoperatively, acute post-operative pain, rescue medication and the incidence of neuropathic pain at 3, 6,12 months postoperatively, also the quality of life measured by EQ-5D questionnaire, adverse events associated with postoperative analgesia.

This study will be conducted under the supervision of an independent auditor. Every week, the auditor checked the data of the participants the day after the surgery was conducted. Assessment of pain intensity and prognostic outcomes must be confirmed by the auditor in sample population. When there is disagreement between surgeon and anesthesiologists in evaluating the prognosis of patients, the auditor must solve this disagreement by discussion with evaluators. Data will be double-entered by two statisticians with limitation of access and locked during statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of inguinal hernia and will receive open inguinal hernia repair (UHS mesh)
* men or woman and 18 ~ 80 years old

Exclusion Criteria:

* body mass index≤18 or≥35
* American Society of Anesthesiology (ASA) classification of anesthesia risk IV and V grade
* allergic to local anesthetics
* hepatic or renal failure
* being pregnant
* skin infection at the puncture site
* pre-operative opioid or non-steroidal anti-inflammatory drugs treatment for chronic pain
* addicted to drugs or alcohol
* uncontrolled general infection
* femoral hernia, incisional hernia or other special types of hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
chronic post-surgical pain | 3 months postoperatively
  chronic post-surgical pain will be measured by visual analogue scale (VAS)

SECONDARY OUTCOMES:
acute post-operative pain | 24h, 48h postoperatively and at discharging time
  pain will be measured by visual analogue scale (VAS)
analgesia rescue | post-operative day 1 to 3
  the dosages of opioid or non-opioid analgesic rescue medication
The incidence of neuropathic pain | 3,6,12 months postoperatively
  the neuropathic pain will be measured by DN4 questionnaire
adverse events | post-operative day 1 to 3
  adverse events related to analgesia: incomplete analgesia; respiratory depression; over-sedation; nausea and vomiting; local hematoma; local infection; muscle weakness; urinary retention
quality of life | 3,6,12 months postoperatively
  the quality of life of patients will be measured by EQ-5D questionnaire
moderate-severe pain | 3,6,12 months postoperatively
  pain will be measured by visual analogue scale (VAS)
chronic post-surgical pain | 6 and 12 months postoperatively
  chronic post-surgical pain will be measured by visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the first affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Crombie IK, Davies HT, Macrae WA. Cut and thrust: antecedent surgery and trauma among patients attending a chronic pain clinic. Pain. 1998 May;76(1-2):167-71. PMID 9696470
- [Background] Martinez V, Baudic S, Fletcher D. [Chronic postsurgical pain]. Ann Fr Anesth Reanim. 2013 Jun;32(6):422-35. doi: 10.1016/j.annfar.2013.04.012. Epub 2013 Jun 7. French. PMID 23747211
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Maia Costa Cabral D, Sawaya Botelho Bracher E, Dylese Prescatan Depintor J, Eluf-Neto J. Chronic pain prevalence and associated factors in a segment of the population of Sao Paulo City. J Pain. 2014 Nov;15(11):1081-1091. doi: 10.1016/j.jpain.2014.07.001. Epub 2014 Jul 16. PMID 25038400
- [Background] Boyers D, McNamee P, Clarke A, Jones D, Martin D, Schofield P, Smith BH. Cost-effectiveness of self-management methods for the treatment of chronic pain in an aging adult population: a systematic review of the literature. Clin J Pain. 2013 Apr;29(4):366-75. doi: 10.1097/AJP.0b013e318250f539. PMID 23042472
- [Background] Werner MU. Management of persistent postsurgical inguinal pain. Langenbecks Arch Surg. 2014 Jun;399(5):559-69. doi: 10.1007/s00423-014-1211-9. Epub 2014 May 23. PMID 24849039
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Galvez R, Marsal C, Vidal J, Ruiz M, Rejas J. Cross-sectional evaluation of patient functioning and health-related quality of life in patients with neuropathic pain under standard care conditions. Eur J Pain. 2007 Apr;11(3):244-55. doi: 10.1016/j.ejpain.2006.02.002. Epub 2006 Mar 24. PMID 16563819
- [Background] Jiang J, Teng Y, Fan Z, Khan MS, Cui Z, Xia Y. The efficacy of periarticular multimodal drug injection for postoperative pain management in total knee or hip arthroplasty. J Arthroplasty. 2013 Dec;28(10):1882-7. doi: 10.1016/j.arth.2013.06.031. Epub 2013 Aug 1. PMID 23910819
- [Background] Alavi SM, Ghoreishi SM, Chitsazan M, Ghandi I, Fard AJ, Hosseini SS, Mahjoobifard M, Fani K. Patient-controlled analgesia after coronary bypass: Remifentanil or sufentanil? Asian Cardiovasc Thorac Ann. 2014 Jul;22(6):694-9. doi: 10.1177/0218492313507783. Epub 2013 Nov 18. PMID 24887897
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Poobalan AS, Bruce J, Smith WC, King PM, Krukowski ZH, Chambers WA. A review of chronic pain after inguinal herniorrhaphy. Clin J Pain. 2003 Jan-Feb;19(1):48-54. doi: 10.1097/00002508-200301000-00006. PMID 12514456
- [Background] Reinpold WM, Nehls J, Eggert A. Nerve management and chronic pain after open inguinal hernia repair: a prospective two phase study. Ann Surg. 2011 Jul;254(1):163-8. doi: 10.1097/SLA.0b013e31821d4a2d. PMID 21562403
- [Background] Lichtenstein IL, Shulman AG, Amid PK, Montllor MM. The tension-free hernioplasty. Am J Surg. 1989 Feb;157(2):188-93. doi: 10.1016/0002-9610(89)90526-6. PMID 2916733
- [Background] van Veen RN, Wijsmuller AR, Vrijland WW, Hop WC, Lange JF, Jeekel J. Long-term follow-up of a randomized clinical trial of non-mesh versus mesh repair of primary inguinal hernia. Br J Surg. 2007 Apr;94(4):506-10. doi: 10.1002/bjs.5627. PMID 17279491
- [Background] Amid PK. The Lichtenstein repair in 2002: an overview of causes of recurrence after Lichtenstein tension-free hernioplasty. Hernia. 2003 Mar;7(1):13-6. doi: 10.1007/s10029-002-0088-7. Epub 2002 Oct 5. PMID 12612791
- [Background] Massaron S, Bona S, Fumagalli U, Battafarano F, Elmore U, Rosati R. Analysis of post-surgical pain after inguinal hernia repair: a prospective study of 1,440 operations. Hernia. 2007 Dec;11(6):517-25. doi: 10.1007/s10029-007-0267-7. Epub 2007 Jul 24. PMID 17646895
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2009 Aug;13(4):343-403. doi: 10.1007/s10029-009-0529-7. Epub 2009 Jul 28. PMID 19636493
- [Background] Miserez M, Peeters E, Aufenacker T, Bouillot JL, Campanelli G, Conze J, Fortelny R, Heikkinen T, Jorgensen LN, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Simons MP. Update with level 1 studies of the European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2014 Apr;18(2):151-63. doi: 10.1007/s10029-014-1236-6. Epub 2014 Mar 20. PMID 24647885
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144